CLINICAL TRIAL: NCT02623010
Title: Phase 2 Study of the Bruton's Tyrosine Kinase Inhibitor Ibrutinib as Maintenance Treatment in Elderly Patients With Primary CNS Lymphoma Following First Line Chemotherapy Treatment
Brief Title: Bruton's Tyrosine Kinase Inhibitor Ibrutinib as Maintenance Treatment in Elderly Patients With Primary CNS Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Osnat Bairey, MD, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0356-15-RMC
Record Dates: First submitted 2015-10-14; First posted 2015-12-07 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Central Nervous System Lymphoma
Keywords: Primary CNS lymphoma; Ibrutinib; Elderly; Maintenance
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Imbruvica (ibrutinib) will be given as maintenance treatment until relapse or toxicity to 30 elderly PCNSL patients after achieving response to first line treatment
  Interventions: Drug: Imbruvica

INTERVENTIONS:
Drug: Imbruvica — Bruton's Tyrosine Kinase Inhibitor Ibrutinib as maintenance treatment in elderly patients with primary CNS lymphoma following first line chemotherapy treatment
  Other Names: Ibrutinib; JNJ-54179060

SUMMARY:
The study will include 30 elderly patients age 60-85 with primary CNS DLBCL . Induction treatment will include Rituximab and high dose methotrexate protocol (containing at least methotrexate and one more chemotherapy agent).

Patients with MRI documented response CR or PR will enter the study protocol maintenance phase which will include continous treatment with Ibrutinib 560 mg day until relapse or disease progression or occurrence of limiting toxicities

DETAILED DESCRIPTION:
30 elderly patients age 60-85 with primary CNS DLBCL who will achieve response CR or PR will enter the study protocol maintenance phase.

Induction treatment will include Rituximab and high dose methotrexate protocol (containing at least methotrexate and one more chemotherapy agent).

Patients with MRI documented response CR or PR will enter the study protocol maintenance phase.

Maintenance: 28 day cycles of Ibrutinib 560 mg orally once daily until relapse or disease progression or occurrence of limiting toxicities

Evaluation of response:

Radiologic evaluation by MRI will be performed every 3 months. Neurologic status evaluation every 2 months Neurocognitive evaluation every 6 months

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed PCNSL patients whose age is >60 years and achieved response (CR/PR) after first line immunochemotherapy treatment
* Tissue diagnosis is mandatory unless positive cerebrospinal fluid (CSF) cytology or vitrectomy are diagnostic with no evidence for systemic disease
* No contraindication for high dose methotrexate (HD-MTX) (adequate renal function)
* KPS > 40%, ECOG < 3
* Hematology values must be within the following limits:

Absolute neutrophil count (ANC) ≥ 1000/µl independent of growth factor support Platelets ≥100,000/µl or ≥50,000/µl if bone marrow involvement independent of transfusion support in either situation • Biochemical values within the following limits: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN) Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft Gault≥ 40 mL/min

-

Exclusion Criteria:

* Major surgery within 4 weeks of randomization.
* History of stroke or intracranial hemorrhage within 6 months prior to randomization.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon).
* Requires treatment with strong CYP3A inhibitors.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
PFS- progression free survival | 3 years
  Progression free survival

SECONDARY OUTCOMES:
Overall survival | 4 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Osnat Bairey, MD, Principal Investigator — Senior Hematologist, Rabin Medical Center
Locations (1):
- Hematology Institute, Petah Tikva, Israel

REFERENCES:
- [Derived] Bairey O, Taliansky A, Glik A, Amiel A, Yust-Katz S, Gurion R, Zektser M, Porges T, Sarid N, Horowitz NA, Shina TT, Lebel E, Cohen A, Geiger KR, Raanani P, Wolach O, Siegal T. A phase 2 study of ibrutinib maintenance following first-line high-dose methotrexate-based chemotherapy for elderly patients with primary central nervous system lymphoma. Cancer. 2023 Dec 15;129(24):3905-3914. doi: 10.1002/cncr.34985. Epub 2023 Aug 12. PMID 37572086